CLINICAL TRIAL: NCT05229562
Title: An Open-Label, Parallel-Group, Phase 1 Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of BIIB122 in Healthy Adult Japanese, Chinese, and Caucasian Participants
Brief Title: A Study to See How BIIB122 Works in the Human Body, and to Evaluate it's Safety, and Tolerability in Healthy Adult Japanese, Chinese, and Caucasian Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 283HV101
Record Dates: First submitted 2022-01-28; First posted 2022-02-08 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — DNL151

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: Low-Dose (Experimental): Participants will receive Dose 1 of BIIB122, orally, once on Day 1.
  Interventions: Drug: BIIB122
- Cohort 2: Mid-Dose (Experimental): Participants will receive Dose 2 of BIIB122, orally, once on Day 1.
  Interventions: Drug: BIIB122
- Cohort 3: High-Dose (Experimental): Participants will receive Dose 3 of BIIB122, orally, once on Day 1.
  Interventions: Drug: BIIB122
- Cohort 4: High-Multi-Dose (Experimental): Participants will receive Dose 3 of BIIB122, orally, once daily (QD), for 10 days.
  Interventions: Drug: BIIB122

INTERVENTIONS:
Drug: BIIB122 — Administered as specified in the treatment arm.
  Other Names: DNL151

SUMMARY:
The study will be looking at an investigational drug, BIIB122, in healthy adult Japanese, Chinese, and Caucasian participants. The main goal of the study is to compare the drug level achieved in the body, between the different ethnic groups, after single and multiple doses of BIIB122. Researchers also want to see if single and multiple doses of BIIB122 are safe and if healthy participants can tolerate given doses of BIIB122.

ELIGIBILITY:
Key Inclusion Criteria:

* Have a body mass index (BMI) between 18 and 30 kilograms per square meter (kg/m^2), inclusive. Body weight (BW) ≥50 kg and ≤100 kg at Screening
* Negative polymerase chain reaction (PCR) test result for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) at Screening and Day -1
* For Japanese healthy volunteers: Participant was born in Japan, and biological parents and grandparents were of Japanese origin; if living outside of Japan for more than 10 years, must not have significantly modified diet since leaving Japan
* For Chinese healthy volunteers: Participant was born in China, and biological parents and grandparents were of Chinese origin; if living outside of China for more than 5 years, must not have had a significantly modified diet since leaving China. Additionally, Chinese healthy volunteers must be of the same gender and have a screening weight within ±15% of their matched Caucasian healthy volunteer
* For Caucasian healthy volunteers: Participant must be a white person of European descent, which may include participants of Hispanic descent. Additionally, Caucasian healthy volunteers must be of the same gender and have a screening weight within ±15% of their matched Japanese healthy volunteer

Key Exclusion Criteria:

* History of any clinically significant cardiac, endocrinologic, hematologic, hepatic, immunologic, infectious, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, and renal, or other major disease, as determined by the Investigator
* History of severe allergic or anaphylactic reactions, or of any allergic reactions that in the opinion of the Investigator are likely to be exacerbated by any component of the study treatment
* Current enrollment in any other drug, biological, device, or clinical study, or treatment with an investigational drug or approved therapy for investigational use within 30 days prior to Day -1, or 5 half-lives, whichever is longer
* Immunization or vaccinations are not allowed from Screening to safety follow-up (SFU)/ early termination (ET) Visit

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2022-09-07 (Actual); Study Completion 2022-09-07 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of BIIB122 | Cohorts 1,2 and 3: At multiple time points post-dose on Days 1 to 4, and at Day 10; Cohort 4: At multiple time points post-dose on Day 1, Pre-dose on Days 2 to 9, Pre-dose and at multiple time points post-dose on Days 10 to 13, and at Day 20
Time to Reach Maximum Observed Plasma Concentration (Tmax) of BIIB122 | Cohorts 1,2 and 3: At multiple time points post-dose on Days 1 to 4, and at Day 10; Cohort 4: At multiple time points post-dose on Day 1, Pre-dose on Days 2 to 9, Pre-dose and at multiple time points post-dose on Days 10 to 13, and at Day 20
Area Under the Concentration-Time Curve From Time 0 to 24 Hours (AUC0-24h) of BIIB122 | Cohorts 1,2 and 3: At multiple time points post-dose on Days 1 to 4, and at Day 10; Cohort 4: At multiple time points post-dose on Day 1, Pre-dose on Days 2 to 9, Pre-dose and at multiple time points post-dose on Days 10 to 13, and at Day 20
Cohorts 1,2 and 3: Area Under the Concentration-Time Curve From Time 0 to Time of the Last Measurable Concentration (AUClast) of BIIB122 | Cohorts 1,2 and 3: At multiple time points post-dose on Days 1 to 4, and at Day 10
Cohorts 1,2 and 3: Area Under the Concentration-Time Curve From Time 0 to Infinity (AUCinf) of BIIB122 | Cohorts 1, 2 and 3: At multiple time points post-dose on Days 1 to 4, and at Day 10
Cohort 4: Cmax of BIIB122 at Steady State (Cmax,ss) | Cohort 4: Pre-dose and at multiple time points post-dose on Days 10 to 13
Cohort 4: Tmax of BIIB122 at Steady State (Tmax,ss) | Cohort 4: Pre-dose and at multiple time points post-dose on Days 10 to 13
Cohort 4: AUC of BIIB122 Within a Dosing Interval at Steady State (AUCtau,ss) | Cohort 4: Pre-dose and at multiple time points post-dose on Days 10 to 13
Cohort 4: Accumulation Ratio (AR) for AUC Within a Dosing Interval (AUCtau) | Cohort 4: Pre-dose and at multiple time points post-dose on Days 10 to 13
Cohort 4: AR for Cmax | Cohort 4: Pre-dose and at multiple time points post-dose on Days 10 to 13

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Cohorts 1,2 and 3: Up to Day 10; Cohort 4: Up to Day 20
  An AE is any untoward medical occurrence in a participant or clinical investigation participant (healthy volunteer) administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. An SAE is any untoward medical occurrence that at any dose results in death, in the view of the investigator, places the participant at immediate risk of death (a life-threatening event), requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, results in a congenital anomaly/birth defect or is a medically important event.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Anaheim Clinical Trials, LLC, Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org